CLINICAL TRIAL: NCT06144983
Title: Chlorhexidine Gel Versus Alvogyl Following Surgical Extraction of Impacted Mandibular Third Molar (Comparative Study)
Brief Title: Chlorhexidine Gel Versus Alvogyl Following Surgical Extraction of Impacted Mandibular Third Molar
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Abdul Haleem Alaa Abdul Zahra, B.D.S, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 417121
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Impacted Third Molar Tooth
Keywords: chlorhexidine gel; Impacted Third Molar Tooth; alvogyl paste
MeSH Terms: interventions — butyl aminobenzoate, eugenol, iodoform, spearmint oil drug combinations; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Alvogyl paste (Experimental): Application of 0.2 gm of Alvogyl paste inside the extraction socket filling it entirely, and suturing the flap interrupted suture following impacted mandibular third molar surgery.
  Interventions: Drug: Alvogyl
- Cholrhexidine gel (Experimental): Application of 1 ml of Chlorhexidine gel inside the extraction socket filling it entirely, and suturing the flap interrupted suture following impacted mandibular third molar surgery.
  Interventions: Drug: Chlorhexidine Gluconate
- control (No Intervention): no dressing material was applied following the impacted mandibular third molar surgery.

INTERVENTIONS:
Drug: Alvogyl — In the first study group, (0.2gm) of Alvogyl paste (Septodont Inc., France), was inserted inside the alveolus, filling it entirely
  Other Names: Alvogyl paste
  Arms: Alvogyl paste
Drug: Chlorhexidine Gluconate — in the second group (1ml) of Periokin (Kin Inc., Spain), containing 0.2% Chlorhexidine bioadhesive gel was injected to fill the entire socket
  Other Names: 0.2% Chlorhexidine gel
  Arms: Cholrhexidine gel

SUMMARY:
Background: One of the most frequent surgical operations in dentistry is the surgical extraction of the impacted mandibular third molar, which is accompanied by a sequelae of swelling, trismus, and pain. Various techniques have been employed to either prevent or reduce these postoperative outcomes.

To the best of our knowledge, few clinical researchers have investigated the effect of local application of Alvogyl paste and Chlorhexidine gel, in the management of pain, facial swelling, and trismus resulting from lower third molar surgical extraction.

Aim of the study: The study was meant to compare the effects of 0.2% chlorhexidine gel and Alvogyl paste on the reduction of the inflammatory reaction caused by the surgical extraction of the impacted mandibular third molar, which includes pain, facial swelling, and trismus.

DETAILED DESCRIPTION:
Background: One of the most frequent surgical operations in dentistry is the surgical extraction of the impacted mandibular third molar, which is accompanied by a sequelae of swelling, trismus, and pain. Various techniques have been employed to either prevent or reduce these postoperative outcomes.

Aim of the study: The study was meant to compare the effects of 0.2% chlorhexidine gel and Alvogyl paste on the reduction of the inflammatory reaction caused by the surgical extraction of the impacted mandibular third molar, which includes pain, facial swelling, and trismus.

Materials and Methods: This randomized control study was conducted from February 2022 to September 2022 on (51) patients, (23) male and (28) female, aged (18-39) years, who presented with impacted mandibular third molar. The participants were randomly allocated into three groups, 17 patients received Alvogyl paste (G1), 17 patients received 0.2% Chlorhexidine gel (Periokin) (G2), and 17 patients received nothing upon surgery (G3). The mouth opening and facial measurements were assessed preoperatively as a baseline reference and on the 2nd and 7th postoperative days. pain was assessed daily using a numerical rating scale (NRS) from the first day to the seventh day following surgery.

Results: Regarding the mouth opening, there was no statistically significant difference among the three groups in the degree of trismus on the second and seventh postoperative days (P ≥ 0.05).

In regards to postoperative facial edema and pain, there was a statistically significant difference among all groups (P < 0.05), however, there was no statistically significant difference between the two study groups.

Conclusion: This study showed that Alvogyl paste and 0.2% Chlorhexidine bioadhesive gel significantly reduce postoperative pain and facial swelling with no significant effect on trismus following impacted mandibular third molar surgical extraction.

ELIGIBILITY:
Inclusion Criteria:

1. Absence of any history of systemic diseases that can impede wound healing or surgical operation.
2. No history of recently using anti-inflammatory drugs.
3. Patients aged ≥18 years who were indicated for surgical extraction of mesioangular, class I or II, and position A or B impacted mandibular third molar.
4. Well-educated patients who had no objection to take part in the study and likely to comply with all study procedures.

Exclusion Criteria:

1. Medical conditions that forbid surgical involvement, such as those in patients with bleeding-related conditions, recent myocardial infarctions, psychological issues, uncontrolled systemic diseases, immune-compromised patients, and patients who were on corticosteroid anti-inflammatory drugs.
2. Recent history of head and neck radiotherapy.
3. Pregnancy, and female patients taking contraceptives.
4. Patients with severe localized infections in relation to the third molar, such as Pericoronitis, or those with severe periodontal disease and/or poor oral hygiene.
5. Patients who were unable to come back for follow-up and recall appointments.
6. Impacted third molar that interferes with the inferior alveolar nerve.
7. Periapical pathology or cystic lesions related to the impacted tooth.
8. Heavy smokers (more than 20 cigarettes/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
postoperative trismus | preoperativly and in the second and seventh postoperative day
  A traditional Vernia caliper is used to measure the distance between the incisal edges of the upper and lower central incisors
postoperative swelling | preoperativly and in the second and seventh postoperative day
  Facial edema was assessed by measuring the distances between three selected lines, utilizing measuring tape, including the tragus of the ear to the outer corner of the mouth, the tragus to the soft tissue pogonion, and the distance that exists between the outer canthus of the eye and the angle of the mandible.
postoperative pain | throughout the first postoperative week
  The intensity of pain was assessed using the numeric rating scale (NRS), on which extreme scores start from zero (no pain) to 10 (worst pain possible). The recording of the pain was on two occasions, one at 10 o'clock am and the other at 10 o'clock pm at the same time except for the operation day in which the first recording was 4 hours after surgery and the second was at 10 o'clock pm, the mean of two records represented the pain for that day.
  The pain was recorded from the day of the operation until the seventh day. The scale was explained to every patient clearly as (0) represents the absence of pain, (1-2) simple pain, (3-4) low pain, (5-6) moderate tolerable pain, (7-8) intolerable severe pain that can be relieved by medication, and (9-10) intolerable severe pain not relieved by medication.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar sh Aladili, B.D.S.MS.C, Study Director — University of Baghdad
Locations (1):
- University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jesudasan JS, Wahab PU, Sekhar MR. Effectiveness of 0.2% chlorhexidine gel and a eugenol-based paste on postoperative alveolar osteitis in patients having third molars extracted: a randomised controlled clinical trial. Br J Oral Maxillofac Surg. 2015 Nov;53(9):826-30. doi: 10.1016/j.bjoms.2015.06.022. Epub 2015 Jul 16. PMID 26188932